CLINICAL TRIAL: NCT06969365
Title: Do Weighted Blankets Reduce Pain and Anxiety Associated With Gynecological Procedures?
Brief Title: Weighted Blankets for IUD Insertion
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Saint Luke's Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SLHS-24-088
Record Dates: First submitted 2025-04-23; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Intra-uterine Device Placement
Keywords: weighted blanket; gynecological procedure; IUD; anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weighted blanket (Experimental): A weighted blanket will be applied to the patient during IUD placement
  Interventions: Other: 10-pound weighted lap-pad
- Non-weighted blanket (Sham Comparator): A non-weighted light blanket will be applied to patient during IUD insertion
  Interventions: Other: blanket

INTERVENTIONS:
Other: 10-pound weighted lap-pad — 10-pound weighted lap pad will be placed over the patient's chest and shoulders
  Arms: Weighted blanket
Other: blanket — A simple, unweighted blanket will be applied to patients during IUD insertion
  Arms: Non-weighted blanket

SUMMARY:
When having an intrauterine device placed in an outpatient clinic, patients frequently feel anxiety related to the procedure. This study is designed to determine if the use of a small, weighted blanket, placed over the patient's chest and shoulders, would help decrease that anxiety, as well as pain related to the procedure.

DETAILED DESCRIPTION:
Patients scheduled for an IUD placement in this specific outpatient clinic will be approached by the study nurse to gauge interest in participating. Consented patients will be randomized to either receive a weighted blanket or a non-weighted blanket. Patients will rate their anxiety on a 100 mm visual-analog scale and pain on a 0-10 verbal scale.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for IUD placement
* age 18 years or older
* able to read and understand English and use a pen

Exclusion Criteria:

* inability to consent
* inability to remove weighted blanket

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale - Anxiety | At the conclusion of the procedure
  Patients will make a mark on a 100 mm line to indicate level of anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Anna Guastello, BSN, Principal Investigator — Saint Luke's Health System
Locations (1):
- Saint Luke's Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nguyen L, Lamarche L, Lennox R, Ramdyal A, Patel T, Black M, Mangin D. Strategies to Mitigate Anxiety and Pain in Intrauterine Device Insertion: A Systematic Review. J Obstet Gynaecol Can. 2020 Sep;42(9):1138-1146.e2. doi: 10.1016/j.jogc.2019.09.014. Epub 2019 Dec 25. PMID 31882291